CLINICAL TRIAL: NCT06702007
Title: eHaRT-A: Adapting an Evidence-based, In-person Harm Reduction Treatment Into a Virtual Care Telehealth Intervention for People With Lived Experience of Homelessness and Alcohol Use Disorder
Brief Title: Electronic Harm Reduction Treatment for Alcohol
Acronym: eHaRT-A
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Tessa Frohe, Assistant Professor, Department of Psychiatry & Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00015865; K01AA030053-02 (NIH)
Record Dates: First submitted 2024-11-19; First posted 2024-11-22 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Alcohol Use Disorder; Harm Reduction; Housing First (eg. Permanent Supportive Housing)
Keywords: Telehealth; Alcohol-Related Harm; Community Based Participatory Research; Lived experience of chronic homelessness
MeSH Terms: conditions — Alcoholism; Harm Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Housing First As Usual (No Intervention): Housing First as usual includes housing provision and management, fulfillment of basic needs (e.g., food, clothing), nursing/medical services and case management.
- Housing First + eHaRT-A (Experimental): HaRT-A comprises three concrete treatment components: 1) measurement and participant-led tracking of indicators of alcohol-related harm (e.g., number of drinks, blackouts), 2) elicitation of harm-reduction and health related quality of life (HRQoL) goals (e.g., drink slower, eat healthier, reconnect with family), and 3) discussion of safer-drinking strategies (e.g., taking B-complex vitamins, eating prior to or during alcohol use, avoiding mixing alcohol and other drugs). HaRT-A honors community representation within harm-reduction intervention development and acknowledges the larger forces (familial, community, geopolitical) at play in substance use, thus emphasizing the wisdom of the participant in defining their own pathway to recovery.
  Interventions: Behavioral: eHaRT-A

INTERVENTIONS:
Behavioral: eHaRT-A — Adaptation of the Harm Reduction Treatment for Alcohol (HaRT-A) into a digital telehealth platform facilitating harm reduction treatment via patient-provider video sessions (eHaRT-A). eHaRT-A will include the three treatment components from the efficacious HaRT-A. eHaRT-A will be delivered during one-on-one sessions through video conferencing with interactive features (i.e., personalized feedback tracked over time and screen sharing).
  Arms: Housing First + eHaRT-A

SUMMARY:
The goal of this project is to transform a successful, face-to-face harm-reduction treatment (HaRT-A) into a digital format, creating eHaRT-A. This new platform is specifically designed for people who have experienced homelessness and an alcohol use disorder (AUD), living within the framework of permanent, supportive, Housing First (HF) facilities. We hypothesize eHaRT-A will be more effective than the standard HF services in reducing alcohol-related harm and improving the overall quality of life for participants.

DETAILED DESCRIPTION:
Brief Summary The goal of this two phased project is to adapt an in-person harm reduction intervention (HaRT-A) into a telehealth platform (eHaRT-A; Phase 1) and test it among individuals with lived experience of homelessness and alcohol use disorder (AUD) in a Housing First (HF) framework (Phase 2). The proposed study will utilize nuanced methodologies that combine community-based participatory research (CBPR) with user-centered technology design. eHaRT-A will be collaboratively adapted with input from HF stakeholders to maximize its acceptability, feasibility, and usability within the HF framework to optimize effectiveness of the eHaRT-A intervention.

Study Design People experiencing homelessness are disproportionately affected by alcohol-related morbidity and mortality with 7 times higher prevalence of AUD than the general population. Traditionally, people with AUD could not attain permanent supportive housing until they attended treatment and achieved abstinence. These requirements served as barriers to housing attainment, relegating people who were not ready, willing or able to stop drinking to continued homelessness. Alternatively, over the past thirty years nonabstinence-based supportive housing, known as Housing First (HF), has emerged as a more effective option by providing immediate, permanent, low-barrier housing to individuals regardless of their alcohol use. HF facilities provide supportive services through HF partners which includes outreach, case management, nursing/medical care, access to external service providers, assistance meeting basic needs [i.e., food, clothing, income, housing]. The HF framework has shown promising effects where those in HF utilized fewer public services (i.e. hospitalizations and emergency service use; jail, and public detoxiﬁcation and sobering center visits), resulting in a nearly four-million-dollar savings to the city of Seattle (in one year) compared to individuals experiencing homelessness who did not access HF resources. Although these ﬁndings are promising, individuals living in HF facilities still report contraindicated levels of drinking and experience signiﬁcant alcohol-related problems. In order to address this need, an in-person, patient-driven, harm-reduction treatment for alcohol (HaRT-A; R34AA022077; PI: Collins) intervention was codeveloped and empirically tested in a randomized controlled trial (RCT). HaRT-A uses a compassionate, non-judgmental, and advocacy-oriented approach. It does not require abstinence or use reduction and comprises 3 treatment components: 1) measurement and participant-led tracking of indicators of alcohol-related harm (e.g., number of drinks, blackouts); 2) elicitation of harm-reduction and health related (HRQoL) goals (e.g., drink slower, eat healthier, reconnect with family); and 3) discussion of safer-drinking strategies (e.g., taking B-complex vitamins, eating prior to or during alcohol use, avoiding mixing alcohol and other drugs). HaRT-A honors community representation within harm-reduction intervention development (ref. 87,88) and acknowledges the larger forces (familial, community, geopolitical) at play in substance use (ref. 89,90), thus emphasizing the wisdom of the participant in deﬁning their own pathway to recovery. The proposed K01 aims to adapt HaRT-A into a telehealth platform (eHaRT-A) to introduce technology-based alcohol-speciﬁc interventions into a HF framework and test it among individuals with lived experience of homelessness and AUD. This project will occur in two phases: Phase 1 will entail codevelopment and iterative testing of the telehealth platform with community stakeholders (i.e., Housing First residents, management, and staff) to leverage stakeholder ideas to inform and build the eHaRT-A prototype and to make design changes that will improve the usability and likeability of the virtual telehealth platform. The primary outcome for Phase 1 is to co-develop (with the CAB) a prototype for eHaRT-A that is deemed usable, feasible, and acceptable by all HF stakeholders (via System Usability Scale [SUS] and Acceptability of Intervention Measure [AIM]). Dr. Frohe will meet the CAB every other week to codesign eHaRT-A (i.e., ensure usable design; Aim 1) and make iterative design changes to improve the acceptability and feasibility of eHaRT-A (i.e., delivery; Aim 2). In Phase 2 an RCT will be conducted (N=160) to test the effectiveness of the eHaRT-A telehealth intervention compared to services as usual (SAU; supportive services provided through HF partners) in improving alcohol-related outcomes (i.e., peak alcohol use, alcohol-related harm, AUD symptoms, and positive urinary ethyl glucuronide tests) and HRQoL over time (Aim 3). The proposed research aligns with national (NIH; NOT-AA-20-011) health initiatives to integrate technology-based interventions for vulnerable and marginalized communities with pre-existing substance use treatments. If successful, this study will lead to the development of a clinically relevant intervention that is more easily transportable to marginalized community settings because it will be developed for, by, and with the community it aims to serve.

Narrative Study Description The proposed study aims will be to leverage stakeholder ideas to inform and build a usable eHaRT-A prototype (Aim 1) and to make iterative design changes that will improve the acceptability and feasibility of the virtual telehealth platform (Aim 2) in Phase 1. The primary outcome for Phase 1 is to co-develop (with the CAB) a prototype for eHaRT-A that is deemed usable, feasible, and acceptable by all HF stakeholders (via System Usability Scale [SUS] and Acceptability of Intervention Measure [AIM]). Self-report on the SUS (ref 101) will also be collected from the group to examine preliminary usability ratings (e.g., clear content portrayal, easy to follow) to evaluate the functionality of eHaRT-A with CAB members in order to enrich and enhance the delivery of eHaRT-A. Based on previous work, a mean score among CAB members of 5 out of a 7-point scale will be considered favorable for the prototype design. (ref. 14,16,98) Phase 2 will entail a randomized controlled trial (RCT) comparing eHaRT-A to services as usual (SAU; supportive services provided through HF partners). This RCT will be a two-armed effectiveness trial and will assess both conditions at baseline, posttest (immediately following treatment end), 1- and 3-month follow-ups. This RCT will test the effectiveness of the eHaRT-A telehealth intervention compared to services as usual (SAU; supportive services provided through HF partners) in improving alcohol-related outcomes (i.e., peak alcohol use, alcohol-related harm, AUD symptoms, and positive urinary ethyl glucuronide tests) and HRQoL over time (Aim 3).

Participants and Recruitment:

Eligible participants will be adults who (1) are registered clients at one of the HF sites, (2) being at least 21 years of age, and (3) fulﬁlling criteria for a current alcohol use disorder (AUD; based on DSM-V semi-structured interview).

Exclusion criterion are (1) refusal or inability to consent to participation in research; (2) constituting a risk to safety and security of other clients or staff; and (3) enrollment in any related treatment studies (incl. studies by this research team). Ability to consent will be assessed during the information session using the UCSD Brief Assessment of Capacity to Consent (UBACC). This 10-item, 3-point Likert-scale measure ensures participants understand the study protocol, potential risks/beneﬁts and their rights as participants prior to study enrollment.

Participants will be recruited from study ﬂyers that will be posted throughout HF facilities to recruit HF residents. Additionally, HF staff, research staff and CAB members will notify HF residents of the opportunity to participate in the study and/or distribute ﬂyers to individuals. Soon thereafter, research staff will be onsite at various HF facilities in rotation to conduct informational sessions (lasting ~20 minutes) and baseline assessments with interested HF residents. During informational sessions, research staff will explain the study procedures, study participants' rights and informed consent materials. If they agree to participate, written informed consent will be obtained, and participants may elect to complete the baseline assessment or schedule it for a later date (within two weeks).

Assessments:

Phase 1: CAB members will complete self-report on the SUS101 during Step 3 of Phase 1 to examine preliminary usability ratings (e.g., clear content portrayal, easy to follow) and to evaluate the functionality of eHaRT-A with CAB members in order to enrich and enhance the delivery of eHaRT-A for HF residents interested in the intervention. Next, Step 4 of Phase 1 will entail an open trial where HF residents will be invited to participate in a single eHaRT-A session. They will complete self-report questionnaires on acceptability (i.e., the AIM,102 SUS,101), alcohol use, and health related quality of life.

Phase 2: Participants will complete EtG urine sample tests and self-report questionnaires on alcohol use and quality of life at baseline, week 2, week 3 and at their 1- and 3-month follow-up appointments. Semi-structured interviews will be also be recorded at the 1-month follow up to examine open ended responses about participant levels of eHaRT-A comprehension, eﬃcacy, and suggestions for its improvement (via Participant Feedback). (ref. 101,102) Finally, qualitative data analysis of participant satisfaction and suggestions for improvement will be conducted using conventional content analysis,(ref. 121) a methodology that facilitates description of qualitative data through a systematic process of coding and classiﬁcation, will be used to delineate common responses to predetermined categories: subjective reactions to the eHaRT-A; intent to use eHaRT-A principles in the future; and suggestions for improvement which can be disseminated through manuscript publications.

ELIGIBILITY:
Inclusion Criteria:

* Being at least 21 years of age
* Speak English fluently
* Currently a registered client at one of the Housing First sites
* Currently drinking (has used alcohol in the past 2 weeks)
* Meeting criteria for "current" (e.g., past-year) AUD according to the Diagnostic and Statistical Manual of Mental Health Disorders, Fifth Edition (determined as scoring >= 2 on the SCID-5-CV)

Exclusion Criteria:

* Enrollment in any related treatment studies (including studies by this research team)
* Refusal or inability to consent
* Constituting a risk to the safety and security of residents or staff

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in physical and mental-health related quality of life from baseline through 3-month follow-up as measured by the EQ-5D-5L | Baseline through 3-month follow-up
  The EQ-5D-5L is a psychometrically sound, 5-item, 5-point Likert scale measure that comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Its summary score will reflect participants' health-related quality of life (HRQoL) as a primary outcome.
Change in typical and peak alcohol quantity consumed from baseline through 3-month follow-up as assessed by the AQUA. | Baseline through 3-month follow-up
  The Alcohol Quantity and Use Assessment (AQUA) was created by the research team for previous studies with a similar population and will be used to record the quantity of alcohol consumed on participants' heaviest and typical drinking days in the past two weeks. Scores are expressed in number of standard drinks with higher numbers indicating heavier drinking.
Change in alcohol-related harm from baseline through 3-month follow-up as assessed by the SIP-2R. | Baseline to 3-month follow-up
  The Short Inventory of Problems (SIP-2R) is a 15-item, Likert-scale questionnaire that measures social, occupational and psychological alcohol-related problems. The summary score will serve as the alcohol-related problems outcome measure.
Feasibility of eHaRT-A within Housing First | Baseline to 3-month follow-up.
  Feasibility will be assessed as ease of enrollment of participants into the study as well as ability to retain participants during the intervention portion of the study (i.e., percentage screened who expressed interest, qualified, and completed eHaRT-A).

SECONDARY OUTCOMES:
Change in motivation/readiness/importance/confidence to engage in harm reduction from baseline through 3-month follow-up as assessed by the MTC. | Baseline through 3-month follow-up
  MTC rulers will be measured using three, 10-point "readiness rulers" (Center for Substance Abuse Treatment, 1999), which assess participants' readiness for, confidence about, and perception of the importance of changing drinking behavior to reduce its "negative side effects," where 0 = not at all ready/confident/important and 10 = totally ready/confident/ important. Readiness rulers have been shown to be associated with alcohol outcomes and have evinced adequate psychometric properties (Bertholet, Gaume, Faouzi, Daeppen, & Gmel, 2012; Heather, Smailes, & Cassidy, 2008; LaBrie, Shiffman, & Earleywine, 2005; Maisto et al., 2011).
Change in alcohol frequency from baseline through 3-month follow-up as assessed by the ASI. | Baseline through 3-month follow-up
  The Alcohol and Substance-use Frequency Assessment questions were adapted from the Addiction Severity Index and will be used to assess frequency of use of alcohol and other substances as well as route of administration.
Change in biochemical verification of EtG from baseline to 3-month follow-up. | Baseline to 3-month follow-up
  Presence of EtG, a direct metabolite of alcohol (cut-off > 500 ng/ml), which is indicative of heavy alcohol use within the past 3 days, will be used as a primary outcome.

OTHER OUTCOMES:
Change in eHaRT receipt/enactment outcomes from baseline to 1-month follow-up as assessed by the SHaRE form. | Baseline through 1-month follow-up.
  The Safer-drinking and Harm Reduction Efforts (SHaRE) form is an open-ended grid created for use in the harm reduction treatment (HaRT-A) to elicit participant-stated goals and safer-drinking tips. The SHaRE will be administered during the initial eHaRT-A sessions and at the follow-up sessions to record participants' current harm reduction goals and to measure whether participants achieved (yes/no) or made measurable progress (yes/no) towards their previously set harm reduction goals according to participants' and interventionists' assessments. The self-reported use of safer drinking strategies will be discussed and monitored during eHaRT-A sessions using the safer drinking portion of the open-ended SHaRE. Reported use of achievement of goals and safer drinking strategies across the course of the study will be used as an outcome in treatment receipt and enactment analyses.
Change in pain from baseline through 3-month as assessed by the BPI. | Baseline through 3-month follow-up
  BPI-SF: Self-report questionnaire (Cleeland; Mendoza, Mayne, Rublee, & Cleeland, 2006), used to assess the severity of pain and the impact of pain on daily functions. There are 9 items asking participants to rate their worst, least, average, and current pain intensity. They are also asked to list current pain-treatments and their perceived effectiveness. They are given a list of current treatments and their perceived effectiveness, and asked to rate the degree that pain interferes with general activity, mood, walking ability, normal work, relations with other persons, sleep, and enjoyment of life on a 10-point scale.
eHaRT-A participant feedback at follow-up. | 1- or 3- month follow-up.
  The Feedback Form will ascertain participants' feedback regarding the eHaRT-A in the form of semi-structured qualitative prompts. This measure will be delivered at the final treatment appointment or the 3-month follow-up if they don't complete the final treatment appointment.
Change in acceptability, effectiveness, and likelihood to engage in eHaRT-A activities as assessed by Acceptability Rulers. | Baseline through 3-month follow-up
  Anticipated Impact and Acceptability Rulers are 5 single, 10-point, items based on an established measure, assessing participants' expectations for how acceptable, effective, helpful, and hopeful they perceive eHaRT-A activities to be for themselves and others.
Acceptability of the eHaRT-A intervention as assessed by the AIM at posttest. | Week 2
  The Acceptability of Intervention Measure (AIM) is made up of 5-point Likert scale items assessing perceived eHaRT-A approval, appeal, likeability, and welcomeness.

CONTACTS AND LOCATIONS:
Overall Officials: Tessa Frohe, PhD, Principal Investigator — University of Washington
Locations (1):
- Downtown Emergency Service Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
The proposed research involves participants from Housing First programs serving highly vulnerable populations, including those experiencing chronic homelessness and substance use disorders. Historical misuse of data on stigmatized behaviors has caused significant harm, including stigma and misrepresentation in politicized media narratives. Sharing individual participant data (IPD) risks breaching anonymity in tight-knit communities and undermining ethical commitments to community-based participatory research (CBPR), which prioritizes data use for the community's benefit. Given these risks, we do not plan to share IPD beyond the specific aims of this study.

REFERENCES:
- [Background] Collins SE, Duncan MH, Saxon AJ, Taylor EM, Mayberry N, Merrill JO, Hoffmann GE, Clifasefi SL, Ries RK. Combining behavioral harm-reduction treatment and extended-release naltrexone for people experiencing homelessness and alcohol use disorder in the USA: a randomised clinical trial. Lancet Psychiatry. 2021 Apr;8(4):287-300. doi: 10.1016/S2215-0366(20)30489-2. Epub 2021 Mar 10. PMID 33713622
- [Background] Collins SE, Malone DK, Clifasefi SL, Ginzler JA, Garner MD, Burlingham B, Lonczak HS, Dana EA, Kirouac M, Tanzer K, Hobson WG, Marlatt GA, Larimer ME. Project-based Housing First for chronically homeless individuals with alcohol problems: within-subjects analyses of 2-year alcohol trajectories. Am J Public Health. 2012 Mar;102(3):511-9. doi: 10.2105/AJPH.2011.300403. Epub 2012 Jan 19. PMID 22390516
- [Background] Collins SE, Clifasefi SL, Nelson LA, Stanton J, Goldstein SC, Taylor EM, Hoffmann G, King VL, Hatsukami AS, Cunningham ZL, Taylor E, Mayberry N, Malone DK, Jackson TR. Randomized controlled trial of harm reduction treatment for alcohol (HaRT-A) for people experiencing homelessness and alcohol use disorder. Int J Drug Policy. 2019 May;67:24-33. doi: 10.1016/j.drugpo.2019.01.002. Epub 2019 Mar 6. PMID 30851620
- [Background] Tsemberis S, Gulcur L, Nakae M. Housing First, consumer choice, and harm reduction for homeless individuals with a dual diagnosis. Am J Public Health. 2004 Apr;94(4):651-6. doi: 10.2105/ajph.94.4.651. PMID 15054020
- See also: Psychiatry Department Project website — https://psychiatry.uw.edu/project/ehart-a-adapting-an-in-person-harm-reduction-for-alcohol-intervention-into-a-telehealth-platform/
- See also: HaRRT Center Project website — https://depts.washington.edu/harrtlab/projects/